CLINICAL TRIAL: NCT01869608
Title: Can we Screen Type 2 Diabetes on the 2nd Day After Delivery in Women Who Had Gestational Diabetes Mellitus?
Brief Title: Postpartum Screening of Type 2 Diabetes
Acronym: Tot ou tard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Full professor, endocrinologist, researcher, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-005
Record Dates: First submitted 2013-05-15; First posted 2013-06-05 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes
Keywords: postpartum screening; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test; Postpartum Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- postpartum screening (Experimental): Oral glucose tolerance test 2 days post-partum
  Interventions: Procedure: oral glucose tolerance test 2 days post-partum

INTERVENTIONS:
Procedure: oral glucose tolerance test 2 days post-partum — Screening for type 2 diabetes after gestational diabetes mellitus.

SUMMARY:
Gestational diabetes mellitus (GDM) complicates 5 to 30 % of pregnancies. GDM is defined as hyperglycemia with onset or first recognition during pregnancy. Because it is a forerunner of type 2 diabetes mellitus (T2DM), professional associations recommend T2DM postpartum screening (T2DM-pPS) at 6 weeks/6 months post delivery, using a 75g oral glucose tolerance test (OGTT).

However, less than a quarter of these women are screened. This recommendation has failed for multiple reasons; the most important being that busy new mothers must deal with the major inconveniences of returning to a sampling center for a 2h testing session, bringing baby along or paying for a sitter, transportation, parking… A mother-friendly solution is direly needed.

The investigators hypothesize that, in these women, results of an OGTT performed after delivery on the last day of their hospital stay (OGTT-1) will predict results of the recommended OGTT (OGTT-2) at 6 weeks/6 months postpartum.

The main aim of our project is to determine the optimal cut-off value for the 2h glucose result during OGTT-1 in order to predict abnormal glucose tolerance status at OGTT-2 (the gold standard), in the same woman.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45 years;
* Having a positive diagnosis of gestational diabetes mellitus (IADPSG criteria);
* Treated with diet or insulin;
* Have given birth to a child at term; gestational age > 37 weeks;
* Have been followed during her pregnancy by a physician who delivers in CHUS;
* Have signed the consent form.

Exclusion Criteria:

* History of glucose intolerance or diabetes before the pregnancy;
* Have presented another obstetrical pathology during the pregnancy;

  * Severe gestational high blood pressure with proteinuria;
  * Delayed intrauterine development syndrome;
  * Pregnancy with more than a foetus;
  * Drug addiction;
  * Had complications during the delivery such as:
* Moderate to severe postpartum bleeding;
* Surgery in postpartum (curettage, hysterectomy, etc.).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of abnormal glucose tolerance | 12 weeks postpartum
  Oral glucose tolerance test

SECONDARY OUTCOMES:
Patient's satisfaction | 12 weeks post-partum
  Satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Clinical Research Center Étienne-Le Bel of the Sherbrooke University Hospital
Locations (1):
- Clinical Research Center Étienne-Le Bel of the Sherbrooke University Hospital, Sherbrooke, Quebec, Canada